CLINICAL TRIAL: NCT00838526
Title: Randomized Double-Blind Parallel Study of Rabeprazole Extended-Release 50 mg vs. Ranitidine 150 mg for Maintenance of Healed Erosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Rabeprazole Extended-Release 50 mg vs. Ranitidine 150 mg for Maintenance of Healed Erosive Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-G000-305
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal; Reflux; Disease; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Disease | interventions — Rabeprazole; Ranitidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rabeprazole ER
- 2 (Active Comparator)
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Rabeprazole ER — 50 mg capsule, taken orally, once daily for 26 weeks.
  Other Names: Aciphex
  Arms: 1
Drug: Ranitidine — 150 mg capsule, taken orally, twice daily for 26 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of rabeprazole extended release (ER) 50 mg (once daily) versus ranitidine 150 mg (twice daily) in the maintenance of complete healing in subjects with healed erosive gastroesophageal reflux disease (eGERD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, parallel-group study. Subjects who meet all eligibility criteria will be randomly assigned to 1 of 2 treatment groups, RAB ER 50 mg (once daily) or Ranitidine 150 mg (twice daily).

ELIGIBILITY:
Inclusion Criteria:

1. Prior completion of Study E3810-G000-301 or -303. Subjects will need to have healed erosive esophagitis (absence of esophageal mucosal breaks or erosions) confirmed by EGD and sustained resolution of heartburn at Visit 4 or 5 of Study E3810-G000-301 or -303.

Exclusion Criteria:

1. Esophageal motility disorders (achalasia, scleroderma, or esophageal spasm).
2. Barrett's esophagus or esophageal stricture.
3. Use of prescription or non-prescription proton pump inhibitors (PPIs), histamine receptor antagonists (H2RA), antacids, sucralfate, misoprostol, prokinetics or drugs with significant anticholinergic effects throughout the study.
4. Subjects who require chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs), oral steroids (>= 20 mg/day prednisone or equivalent), or aspirin (->; 325 mg/day).
5. Significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities that would be likely to interfere with the conduct of the study, the interpretation of study results, or the health of the subject during the study.
6. Any condition that would make the subject, in the opinion of the investigator or sponsor, unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-08-31 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2009-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rossiter, MD, Study Director — Eisai Inc.
Locations (4):
- United States (4):
  - Ltd., Moline, Illinois
  - Midwest Clinical, Moline, Illinois
  - Research Associates, Moline, Illinois
  - Moline, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible for this study if they had completed one of the healing studies (E3810-G000-301 or E3810-G000-303), had no evidence of oesophageal erosions, had sustained heartburn resolution, and had no record of any serious adverse event (SAE) related to study medication during the healing study.
Pre-assignment Details: Out of the 240 participants who were randomized in this study, 235 participants received study treatment.
Groups:
- RAN 150mg BID: Morning dose included 1 x Placebo to match RAB (Rabeprazole) ER (Extended Release) 50mg capsule and 1 x RAN (Ranitidine) 150mg capsule. Evening dose included 1 x RAN 150mg capsule. Received study drug orally daily for 26 weeks.
- RAB ER 50mg QD: Morning dose included 1 x RAB ER 50mg capsule and 1 x Placebo to match RAN 150mg capsule. Evening dose included 1 x Placebo to match RAN 150mg capsule. Received study drug orally daily for 26 weeks.
Period: Overall Study
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Started | 59 (Treated) | 176 (Treated)
Completed | 35 | 137
Not Completed | 24 | 39
Not completed — Adverse Event | 3 | 12
Not completed — Lost to Follow-up | 4 | 12
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lack of Efficacy | 2 | 3
Not completed — Other | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAN 150mg BID | RAB ER 50mg QD | Total
Number analyzed (Participants) | 59 | 176 | 235
Age, Customized [Mean (Standard Deviation); unit: Years] | 46.7 (12.15) | 46.4 (12.83) | 46.5 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 81 | 108
  Male | 32 | 95 | 127

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Investigator-recorded Sustained Resolution of Heartburn at Week 26
Description: Heartburn or other GERD-associated symptoms (regurgitation, epigastric or chest pain, dysphagia, belching, bloating, early satiety, other) was based on a 4-point Likert scale that included the following: None (No symptoms); Mild (Awareness of symptoms but easily tolerated); Moderate (Discomforting symptom sufficient to cause interference with normal activities including sleep); Severe (Incapacitating symptom, inability to perform normal activities).
Time Frame: Baseline to Week 26
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Number analyzed (Participants) | 59 | 176
Percentage of Participants
  Yes | 8.5 | 57.4
  No | 25.4 | 18.8
  Missing | 66.1 | 23.9

2. Primary Outcome: Percentage of Participants With Maintenance of Complete Healing of eGERD at Week 26
Description: eGERD (erosive gastroesophageal reflux disease) healing measured by the Time-to-Relapse of Oesophageal Erosions using an Esophagogastroduodenoscopy (EGD). Lesions were identified and graded using the following Los Angeles (LA) classification of Oesophagitis: Not Present: No breaks (erosions) in the esophageal mucosa (however, edema, erythema, or friability may be present). Grade A: One or more mucosal breaks not more than 5mm in maximum length. Grade B: One or more mucosal breaks more than 5mm in maximum length, but not continuous between the tops of 2 mucosal folds. Grade C: Mucosal breaks continuous between the tops of 2 or more mucosal folds, but involving less than 75% of the esophageal circumference. Grade D: Mucosal breaks involving at least 75% of the esophageal circumference.
Time Frame: Baseline to Week 26
Population: Intent-to-Treat (ITT) Population - all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Number analyzed (Participants) | 59 | 176
Percentage of Participants | 32.9 | 84.9

3. Secondary Outcome: Percentage of Participants With Adverse Events by Category
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered an investigational product. A treatment emergent AE (TEAE) was any AE beginning on or after the confirmed date of first dose of study medication, up to and including 7 days after the last dose of study medication. A TEAE was considered related to study treatment if a causal relationship between the study treatment and the AE was a reasonable possibility. AEs were graded as severe if they were incapacitating, with inability to work or to perform normal daily activity. Serious AEs (SAEs) were events that resulted in death, were life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or were a congenital anomaly/birth defect.
Time Frame: From the time of administration of the first dose of study drug up to a maximum of approximately 30 weeks.
Population: The safety population included all randomized participants who received at least one dose of study drug and had at least one post-baseline safety assessment. Analyses of the safety population was based on the actual treatment participants received.
Measure: Number; unit: Percentage of participants
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
Number analyzed (Participants) | 59 | 173
Percentage of participants
  Any TEAE | 47.5 | 64.2
  Treatment-related TEAE | 8.5 | 14.5
  Severe TEAE | 3.4 | 8.1
  Severe, treatment-related TEAE | 1.7 | 0.6
  Death | 0 | 0
  Other SAE | 1.7 | 6.4
  Treatment-related SAE | 0 | 0
  TEAEs leading to discontinuation of treatment | 6.8 | 6.9

ADVERSE EVENTS:
Time Frame: From the time of administration of the first dose of study drug up to a maximum of approximately 30 weeks.
Description: Data are presented as number of participants with treatment emergent AEs (serious and non-serious). The analysis was performed using the safety population, defined as all participants who received at least 1 dose of study drug and had a postbaseline safety assessment. All-cause mortality was reported for all participants randomized.
Arm/Group | RAN 150mg BID | RAB ER 50mg QD
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/176
Serious Adverse Events (participants affected / at risk) | 1/59 | 10/173
Other Adverse Events (participants affected / at risk) | 8/59 | 43/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAN 150mg BID (N=59) | RAB ER 50mg QD (N=173)
Angina pectoris (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAN 150mg BID (N=59) | RAB ER 50mg QD (N=173)
Gastritis (Gastrointestinal disorders) | 1 | 13
Sinusitis (Infections and infestations) | 1 | 11
Hiatus hernia (Gastrointestinal disorders) | 2 | 10
Nausea (Gastrointestinal disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No